CLINICAL TRIAL: NCT05391763
Title: Bilateral Prophylactic Mastectomy; Should we Preserve the Pectoral Fascia?: Protocol of a Dutch Double Blinded, Prospective, Randomized Controlled Pilot Study With a Within-subject Design
Brief Title: Bilateral Prophylactic Mastectomy; Should we Preserve the Pectoral Fascia?
Acronym: PROFAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Linetta Koppert, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL72939.078.20; NTR7620 (Registry Identifier: trialregister.nl)
Record Dates: First submitted 2022-05-17; First posted 2022-05-26 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: BRCA1/2 Mutation; Bilateral Prophylactic Mastectomy; Seroma; Pectoral Fascia
MeSH Terms: conditions — Seroma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The patient and the observer for drain volume are both blinded for their assigned breast randomization. The surgeon(s) and coordinating researcher will not be blinded, and are therefore not allowed to measure the drain production.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right: removal of fascia pectoralis, left: preservation of fascia pectoralis (Other)
  Interventions: Procedure: Fascia pectoralis preservation
- Left: removal of fascia pectoralis, right: preservation of fascia pectoralis (Other)
  Interventions: Procedure: Fascia pectoralis preservation

INTERVENTIONS:
Procedure: Fascia pectoralis preservation — A total mastectomy will be performed in the control breast: a procedure which includes removal of the breast glandular tissue including the PF and subcutaneously excision of the nipple-areolar complex, while the pectoralis muscle will be spared. As much of the healthy skin envelope will be preserved to enable the performance of an effective breast reconstruction afterwards. When a nipple-sparing mastectomy is performed, the skin envelope together with the nipple-areolar complex will be spared. The investigational part of the operation is preservation of the PF. Dissection of cutaneous flaps and the breast with or without the PF will be performed with electrocautery.

SUMMARY:
Many surgical guidelines promote the removal of the pectoral fascia in mastectomies for invasive breast cancer, but there is no evidence to support this statement in (bilateral) prophylactic mastectomies. Reported wound-related local complications following mastectomy include seroma, flap necrosis, infection, hematoma, and nerve injury. Seroma causes discomfort and may delay the reconstructive procedures. Whether the removal or preservation of the pectoral fascia influences seroma formation following mastectomy remains unclear to our knowledge.

DETAILED DESCRIPTION:
The primary objective of this pilot study is to investigate the impact of removal versus preservation of the pectoral fascia on drain policy and needle aspirations in women who undergo a bilateral prophylactic mastectomy. The secondary objective is to investigate the impact of removal versus preservation of the pectoral fascia on postoperative (surgical) complications.

The study design includes a double-blinded, prospective, randomized controlled pilot study with a within-subject design. All patients will undergo a bilateral prophylactic mastectomy and randomization will occur within the patient. Preservation of the PF will be performed in one breast (intervention), while removal of the PF will be performed in the contralateral breast of the same patient (control). Consequently, the operation involves a total bilateral prophylactic mastectomy, with unilateral preservation of the PF

The follow-up time of each patient will be 6 weeks. The patients' files will be viewed after the removal of the drain for additional recorded variables.

ELIGIBILITY:
Inclusion Criteria:

* Female patient
* Scheduled for a bilateral prophylactic mastectomy in the Erasmus MC Academic Breast Cancer Centre in Rotterdam
* Ability to give written consent
* Adequate understanding of Dutch language

Exclusion Criteria:

* History of diagnosis of invasive breast cancer or ductal carcinoma in situ (DCIS)
* Other malignancies

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Drainproduction in milliliters | Until drain removal, maximum 1 week
  The total drainage volume of the left and right breast in milliliters
Time to drain removal in days | Until drain removal, maximum 1 week
  Number of days until drain removed

SECONDARY OUTCOMES:
Seroma (yes/no) | Up to 6 weeks
  Occurrence of seroma
Needle aspirations (number) | Up to 6 weeks
  Number of needle aspirations
Postoperative pain (score 1-10) | Up to 6 weeks
  Postoperative pain measured with Visual Analogue Scale
Postoperative bleeding (yes/no) | Up to 6 weeks
  Occurrence of postoperative bleeding
Wound related issues (yes/no) | Up to 6 weeks
  Wound related issues such as hematoma or infection
Hospitalization duration (in days) | Up to 6 weeks
  Duration of hospitalization, including readmissions

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clarijs ME, van Egdom LSE, Verhoef C, Vasilic D, Koppert LB; PROFAS Collaborator Group. Bilateral prophylactic mastectomy: should we preserve the pectoral fascia? Protocol of a Dutch double blinded, prospective, randomised controlled pilot study with a within-subject design (PROFAS). BMJ Open. 2023 Feb 17;13(2):e066728. doi: 10.1136/bmjopen-2022-066728. PMID 36806067